CLINICAL TRIAL: NCT02033642
Title: A Family-Based Weight Loss Intervention for Youth With Intellectual Disability
Acronym: HealthU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Richard Fleming, Professor (retired), University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HealthU R01; 5R01HD072573-03 (NIH)
Record Dates: First submitted 2014-01-03; First posted 2014-01-13 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: weight loss, nutrition, physical activity, lifestyle, intellectual disability, adolescence, families
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity; Intellectual Disability | interventions — Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Based Behavioral Intervention (Experimental): Family Based Behavioral Intervention (FBBI) is a 24-session lifestyle intervention designed to: (1) educate adolescent/young adult participants and their parents in principles of good nutrition and physical activity, and (2) train parents to implement lifestyle changes at home to facilitate weight loss in their child.
  Interventions: Behavioral: Family Based Behavioral Intervention
- Maintenance (Experimental): The Maintenance condition in this study is a 12-session intervention designed to extend FBBI and continue to teach adolescent/young adult participants and their parents to continue practicing lifestyle behaviors at home.
  Interventions: Behavioral: Maintenance

INTERVENTIONS:
Behavioral: Family Based Behavioral Intervention — Family Based Behavioral Intervention (FBBI) is a 24-session lifestyle intervention designed to: (1) educate adolescent/young adult participants and their parents in principles of good nutrition and physical activity, and (2) train parents to implement lifestyle changes at home to facilitate weight loss in their child by monitoring diet and physical activity behaviors, setting goals, providing support and reinforcement, and assessing and making changes to the home environment.
  Arms: Family Based Behavioral Intervention
Behavioral: Maintenance — The Maintenance condition in this study is a 12-session intervention designed to extend FBBI and continue to teach adolescent/young adult participants and their parents to continue practicing lifestyle behaviors, generalize healthful behaviors to new environments, find additional social and community supports, and prevent and manage relapse.
  Arms: Maintenance

SUMMARY:
The purpose of this randomized controlled trial is twofold. First, to examine the efficacy of a 24-session, 6-month family-based behavioral intervention (FBBI) - as compared to a waitlist FBBI group, which later receives the same FBBI - that targets weight loss in adolescents/young adults with intellectual disability aged 14-22 years. Second, to examine the efficacy of a 12-session, 6-month Maintenance intervention that targets maintenance of weight loss in the same population of adolescents/young adults with intellectual disability. The Maintenance condition follows the completion of each FBBI group and involves a re-randomization to either the Maintenance intervention or no further intervention. Primary outcome measures include body weight and Body Mass Index (BMI). Secondary outcome measures include physical activity/sedentary behavior (measured via accelerometry), dietary patterns (3-Day Food Records), and self-efficacy (brief questionnaire). Hypotheses are that: (1) participants in the FBBI condition will lose more weight (and reduced BMI) than participants in the waitlist treatment condition, and that (2) participants in the Maintenance condition will maintain weight lost (and reductions in BMI) or experience less weight regain, as compared with participants who receive no further intervention following FBBI.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria for the adolescents with intellectual disability (ID) will be:

1. Age 14-22 years
2. Clinically overweight or obese, as indicated by BMI guidelines set by the Centers for Disease Control and Prevention
3. Scores of ≤ 75 on the Kaufman Brief Intelligence Test (KBIT) and Vineland Adaptive Behavior Scales, 2nd Edition to establish criteria for the presence of an intellectual disability
4. Living at home in a single- or two-parent family with no plans to leave home in the next year
5. Verbal ability and necessary behavioral/social skills to participate in a group classroom-based educational program (determined by clinical observation and judgment accomplished through a structured interview during enrollment)
6. Signed approval to participate by the adolescent's primary care provider (and by other specialists such as cardiologists or neurologists if the participant has a heart condition or neurological disorder).

Exclusion Criteria: Exclusion criteria will be:

1. Cardiac problems that preclude participation in moderate-to-vigorous-physical-activity (MVPA)
2. Insulin-dependent diabetes
3. An active seizure disorder not stabilized on medication
4. Non-ambulatory, i.e. uses a wheelchair, or orthopedic injuries/deformities that prohibit moderate walking and other exercise
5. Colitis, Crohn's Disease, and Inflammatory Bowel Disease
6. Prader Willi syndrome
7. Unwillingness to wear the accelerometer at screening or enrollment
8. Recent history of disruptive, inappropriate or dangerous behaviors (e.g., self-injury, aggression/injury to others, property destruction, and extreme and ongoing use of inappropriate language).

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2012-08-22 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline (BL), change from BL to 6 months, change from BL to 12 months and change from BL to 18 months
  Adolescent/young adult participants' body weight was measured in kg using a Seca digital scale.
Body Mass Index (BMI) | Baseline (BL), change from BL to 6 months, change from BL to 12 months and change from BL to 18 months
  Adolescent/young adult participants' BMI was determined by taking their height and weight on a Seca digital scale and stadiometer, respectively, and calculating their BMI.

SECONDARY OUTCOMES:
Physical activity | Baseline (BL), change from BL to 6 months, change from BL to 12 months and change from BL to 18 months
  Physical activity refers to participants' physical movement, performed at light, moderate, and vigorous levels of exertion. Physical activity was measured via Actigraph accelerometers worn over 7 day intervals at each measurement point - baseline, 6 months, 12 months and 18 months. In addition to light, moderate and vigorous physical activity, sedentary behavior was also estimated from the Actigraph records.
Dietary patterns | Baseline (BL), change from BL to 6 months, change from BL to 12 months and change from BL to 18 months
  Dietary patterns refers to consistencies in each participants' food intake, determined via analysis of 3-Day Food Records completed at each measurement point: baseline, 6 months, 12 months, and 18 months.
Self-Efficacy | Baseline (BL), change from BL to 6 months, change from BL to 12 months and change from BL to 18 months
  Self-efficacy is a measure of a participant's perceived confidence in their ability to competently engage in a behavior. In this study, self-efficacy is assessed for adolescent participants' dietary and physical activity behaviors. Self-efficacy was obtained via a brief, 2-question interview with the adolescent participants.

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Fleming, PhD, Principal Investigator — University of Massachusetts Boston - retired
Locations (1):
- University of Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curtin C, Bandini LG, Must A, Gleason J, Lividini K, Phillips S, Eliasziw M, Maslin M, Fleming RK. Parent support improves weight loss in adolescents and young adults with Down syndrome. J Pediatr. 2013 Nov;163(5):1402-8.e1. doi: 10.1016/j.jpeds.2013.06.081. Epub 2013 Aug 20. PMID 23968742